CLINICAL TRIAL: NCT06896110
Title: Phase 1 Trial of Intrathecal Azacitidine and Nivolumab in Patients With Recurrent High-grade Glioma
Brief Title: Intrathecal Azacitidine and Nivolumab in Patients With Recurrent High-grade Glioma
Status: Enrolling by invitation | Phase: Phase 1 | Type: Interventional
Sponsor: Andrew P. Groves (Other)
Responsible Party: Sponsor-Investigator, Andrew P. Groves, Clinical Assistant Professor, University of Iowa
Organization: University of Iowa (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 202406429
Record Dates: First submitted 2025-03-19; First posted 2025-03-26 (Actual); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Glioblastoma (GBM); Diffuse Midline Glioma (DMG); Astrocytoma, IDH-Mutant, Grade 4; Diffuse Hemispheric Glioma, H3 G34-Mutant; Gliosarcoma of Brain
MeSH Terms: conditions — Glioblastoma; Astrocytoma | interventions — Nivolumab; Azacitidine; Spinal Puncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (IT nivolumab + IT azacitidine) (Experimental): Patients will receive intrathecal azacitidine on day 1, 8, and 22 of cycle 1 (34 day cycle). Intrathecal nivolumab will be given at a flat dose of 40 mg on day 8 and 22. Each subsequent cycle will be 28 days with intrathecal azacitidine and intrathecal nivolumab given on days 1 and 15. Intrathecal azacitidine will be dose-escalated with 4 dose levels (5, 10, 20, 40 mg) using a 3+3 design. Patients may continue on study in the absence of disease progression or unacceptable toxicity. Patients will have CSF and blood specimen collection on days 1 and 8 of cycle 1, and then day 1 of every-other cycle starting with cycle 2. Patients will undergo MRI at baseline, then every 8 weeks (e.g. after cycle 3, cycle 5, etc…).
  Interventions: Drug: Nivolumab; Drug: Azacitidine (AZA); Procedure: lumbar puncture; Diagnostic Test: MRI Contrast

INTERVENTIONS:
Drug: Nivolumab — Intrathecal nivolumab will be given at a flat dose of 40 mg
Drug: Azacitidine (AZA) — Intrathecal azacitidine will be dose-escalated with 4 dose levels (5, 10, 20, 40 mg) using a 3+3 design.
Procedure: lumbar puncture — Lumbar puncture for intrathecal delivery and collection of CSF
Diagnostic Test: MRI Contrast — MRI Brain and full Spine (with and without contrast) will be performed prior to enrollment. During trial therapy, MRI Brain (with and without contrast) will be performed after cycle 1 and after that every 8 weeks (e.g. after cycle 3, cycle 5, etc…)

SUMMARY:
This is a single-arm open-label phase 1 dose escalation/expansion trial assessing the safety and efficacy of concurrent intrathecal azacitidine and intrathecal nivolumab in recurrent high-grade glioma.

DETAILED DESCRIPTION:
PRIMARY OUTCOME Phase I To determine the safety and maximum tolerated dose (MTD) of intrathecal (IT) azacitidine in combination with IT nivolumab in patients with recurrent high-grade glioma

Expansion Cohort To estimate the overall response rate (ORR)

SECONDARY OUTCOMES

To estimate:

1. Duration of response (DOR)
2. Progression-free survival (PFS)
3. Overall survival (OS)

EXPLORATORY OUTCOMES Changes in immune profiling (flow cytometry, cytokine/chemokine analysis) and circulating tumor DNA (ctDNA) biomarkers (quantification, DNA methylation)

ELIGIBILITY:
INCLUSION CRITERIA

1. For patients age ≥ 18: Able and willing to provide written informed consent
2. For patients aged 13-17: Parent/guardian of adolescent patient must have the ability to provide written informed consent. Adolescent patients must have the ability to provide written informed assent.
3. Stated willingness to comply with all trial procedures and availability for the duration of the trial
4. Histologically confirmed diagnosis of World Health Organization Grade IV high-grade glioma. Eligible diagnoses include: Glioblastoma (IDH-wildtype), Gliosarcoma, Diffuse Midline Glioma (H3 K27-altered), diffuse hemispheric glioma (H3 G34-mutant), diffuse pediatric-type high-grade glioma (H3 and IDH-wildtype), Astrocytoma IDH-mutant (Grade 4)
5. Previous first-line treatment with at least radiotherapy (and temozolomide in the case of glioblastoma or astrocytoma IDH-mutant (grade 4))
6. Documented recurrence by diagnostic biopsy or contrast-enhanced magnetic resonance imaging (MRI) per RANO 2.0 criteria
7. At least one measurable lesion per RANO 2.0 meeting the following criteria: Contrast-enhancing or non-enhancing lesions with clearly defined margins by MRI Scan, with both perpendicular diameters on a single slice of at least 10 mm, visible on two or more slices that are preferably, at most, 3 mm apart with 0-mm interslice gap.
8. Age ≥ 13
9. Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 (age ≥ 16) or Lansky of ≥ 60 (age <16)
10. Disease status confirmed with baseline imaging performed within 28 days of Day 1 of trial treatment. Patients with extracranial metastatic or leptomeningeal disease will be excluded (see Section 5.2)
11. Subjects must be on a stable or decreasing dose of corticosteroids for at least 7 days before enrollment
12. Patients must have organ and marrow function as defined below:

    Eligibility Guidelines of Organ and Marrow Function Hematologic Absolute neutrophil count (ANC) ≥ 1.5 x 109/L Hemoglobin ≥ 9.0 g/dL Platelets ≥ 75 x 109/L PT/INR and PTT ≤ 1.5 X ULN Hepatic Total bilirubin ≤ 1.5 X ULN (except subjects with known Gilbert syndrome, who can have total bilirubin < 3.0 mg/dL AST and ALT ≤ 3.0 X ULN Renal Creatinine OR Calculated creatinine clearance OR 24-hour urine creatinine clearance ≤ 2 X ULN
    * 50 mL/min
    * 50 ml/min
13. Women of childbearing potential (WOCBP) must have a negative serum or urine pregnancy test within 24 hours of starting therapy
14. WOCBP must agree to follow instructions for methods of contraception
15. Men who are sexually active with WOCBP must agree to follow instructions for methods of contraception
16. Investigators will counsel WOCBP and male subjects who are sexually active with WOCBP on the importance of pregnancy prevention and implications of an unexpected pregnancy. At a minimum subjects must agree to the use of two methods of contraception, with one method being highly effective and the other method being either highly effective or less effective: starting at ICF or first dose and continuing 6 months after last dose of trial treatment:

    Highly effective methods of contraception Male condoms with spermicide Hormonal methods including combined oral contraceptive pills, vaginal ring, injectables, implants, and intrauterine devices (IUD) Non-hormonal IUD Tubal ligation Vasectomy Complete Abstinence

    Less effective methods of contraception Diaphragm with spermicide Cervical cap with spermicide Vaginal sponge Male condom without spermicide Progestin only pills Female condom
17. An interval of ≥ 2 weeks from major surgery
18. An interval of ≥ 4 weeks from chemotherapy, radiotherapy, or other investigational agents

EXCLUSION CRITERIA

1. Presence of extracranial metastatic or leptomeningeal disease
2. Patients with diffuse intrinsic pontine glioma, defined as tumors with a pontine epicenter and diffuse involvement of the pons
3. Patients must not have active autoimmune disease that has required systemic treatment in the past 2 years (e.g. use of disease modifying agents, corticosteroids, or immunosuppressive drugs)
4. Prior azacitidine for the treatment of cancer (prior administration of nivolumab or other immune checkpoint inhibitor is allowed)
5. Subjects with major medical, neurologic, or psychiatric condition who are judged to be unable to fully comply with trial therapy or assessments
6. Positive test for hepatitis B or C virus indicating acute or chronic infection, given the risk of reactivation with checkpoint inhibition
7. Known history of testing positive for HIV or known acquired immunodeficiency syndrome (AIDS), due to the unknown effects of HIV on the immune response to intrathecal azacitidine and nivolumab
8. Patients with a history of pneumonitis
9. Evidence of active infection requiring treatment with IV antibiotics ≤ 7 days prior to initiation of trial therapy.
10. History of allergy to trial drug components
11. Prisoners or subjects involuntarily incarcerated

Patients of all genders, races, and ethnicities are invited to participate.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-06-05 (Actual); Primary Completion 2027-03 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events | 24 months
  Adverse events will be graded by the Common Terminology Criteria for Adverse Events version 5.0.
Maximum tolerated dose (MTD) of intrathecal azacitidine in combination with intrathecal nivolumab | 24 months
  The MTD will be established using a 3+3 design.
Overall Response Rate (Expansion Cohort) | 24 months
  The primary objective of the expansion cohort is to obtain a preliminary estimate of the overall response rate (ORR). ORR will be defined as the proportion of patients with a complete response (CR) or partial response (PR) according to Response Assessment in Neuro-Oncology (RANO) 2.0 criteria

SECONDARY OUTCOMES:
To estiamte the duration of response (DOR) | 24 months
  DOR will be defined as the time from first documented complete response (CR) or partial response (PR) to progressive disease (PD) according to RANO 2.0 criteria
To estimate progression-free survival | 24 months
  PFS will be defined as the time from trial treatment initiation to first documented progression or death due to any cause.
To estimate overall survival | 24 months
  OS will be defined as the time from trial treatment initiation to death due to any cause.
To assess biomarkers for immunologic and epigenetic effects of therapy | 24 months
  Changes in CSF and blood immunological profiling by flow cytometry, cytokine/chemokine analysis. Changes in circulating tumor DNA (ctDNA) analysis in CSF

CONTACTS AND LOCATIONS:
Locations (1):
- Holden Comprehensive Cancer Center, Iowa City, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and Informed Consent Form (ICF)
Supporting Information: Study Protocol, ICF